CLINICAL TRIAL: NCT02533375
Title: A Multicenter, Open-Label Study of Adalimumab in Japanese Subjects With Generalized Pustular Psoriasis
Brief Title: Study to Investigate Efficacy and Safety of Adalimumab in Japanese Subjects With Generalized Pustular Psoriasis (GPP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-193
Record Dates: First submitted 2015-08-20; First posted 2015-08-26 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-07

CONDITIONS: Generalized Pustular Psoriasis (GPP); Adalimumab; Japanese
Keywords: efficacy; safety
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving adalimumab (Experimental): 80 mg at Week 0 by subcutaneous (SC) injection, followed by 40 mg every other week (eow) on and after Week 2 until Week 50. Dose escalation to 80 mg eow was allowed for participants who did not have adequate response on or after Week 8.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous injection
  Other Names: Humira; ABT-D2E7

SUMMARY:
The purpose of this study was to investigate the efficacy, safety, and pharmacokinetics of adalimumab in Japanese participants with generalized pustular psoriasis (GPP) who did not have an adequate response to their currently approved treatment.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, open-label, single-arm study of adalimumab in Japanese participants with generalized pustular psoriasis (GPP). The study included a 30-day screening period, a 52-week treatment period, and a 70-day follow-up period. The dose regimen of adalimumab used in this study was 80 mg at Week 0 by subcutaneous (SC) injection, followed by 40 mg every other week (eow) on and after Week 2 until Week 50. Dose escalation to 80 mg eow was allowed for participants who did not have adequate response on or after Week 8.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized pustular psoriasis
* Total skin score of at least 3 and erythema with pustules (skin score of at least 1) at baseline in the Japan Dermatology Association (JDA) severity index of Generalized Pustular Psoriasis (GPP) in GPP Medical Care Guideline 2014 in Japan
* Inadequate response to, or intolerance to, or contraindication to the currently approved GPP treatment (excluding infliximab)
* Infliximab secondary failure, or intolerant to infliximab

Exclusion Criteria:

* Erythrodermic psoriasis, guttate psoriasis or sub-corneal pustular dermatosis at Screening
* Drug-induced GPP
* Cannot stop ongoing use of prohibited GPP treatments
* Total JDA severity index of GPP of 14 or more in GPP Medical Care Guideline 2014 in Japan

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09-28; Primary Completion 2016-09-15 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Robinson, PharmD, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: AbbVie — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Full Analysis Set (FAS) included all participants who received at least 1 dose of study drug and had at least 1 post-treatment efficacy assessment.
Period: Overall Study
Arm/Group | Participants Receiving Adalimumab
Started | 10
Completed | 5
Not Completed | 5
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of study drug and had at least 1 post-treatment efficacy assessment.
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Generalized Pustular Psoriasis (GPP) Duration [Mean (Standard Deviation); unit: years] | 10.6 (12.59)
Prior GPP Therapy [Count of Participants; unit: Participants]
  Psoralen and ultraviolet A light (PUVA) | 1
  Narrow-band ultraviolet B light (UVB) | 2
  Granulocyte and Monocyte Absorbent Apheresis (GMA) | 2
  None of the above | 5
Prior Infliximab Use [Count of Participants; unit: Participants]
  Yes | 3
  No | 7

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving Clinical Response at Week 16
Description: Clinical Response was defined as reduction of the Generalized Pustular Psoriasis (GPP) total skin score (range 0-9, with 9 representing severe symptoms) relative to baseline (Day 1), according to Japan Dermatology Association (JDA) severity index in GPP medical care guideline 2014. The total skin score is the combined skin scores for area of erythema (redness), area of erythema with pustules (small pockets of pus), and area of edema (swelling). Clinical Response was defined as the improvement (reduction) of total skin score of at least 1 point (if the participant's baseline total skin score was 3); improvement (reduction) at least 2 points (if the participant's baseline total skin score was 4-9); or remission if the total skin score was 0.
Time Frame: Baseline and Week 16
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of study drug and had at least 1 post-treatment efficacy assessment; non-responder imputation was used for participants with missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants | 7

2. Secondary Outcome: Number of Participants Achieving Clinical Response Over Time
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 24, Week 36, Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
participants
  Week 2 | 5
  Week 4 | 6
  Week 8 | 6
  Week 12 | 5
  Week 24 | 6
  Week 36 | 6
  Week 52 | 5

3. Secondary Outcome: Number of Participants Achieving Clinical Remission Over Time
Description: The Generalized Pustular Psoriasis (GPP) total skin score (range 0-9, with 9 representing severe symptoms) was calculated according to Japan Dermatology Association (JDA) severity index in GPP medical care guideline 2014. The total skin score is the combined skin scores for area of erythema (redness), area of erythema with pustules (small pockets of pus), and area of edema (swelling). Clinical remission was defined as a total skin score of 0.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
participants
  Week 2 | 0
  Week 4 | 1
  Week 8 | 0
  Week 12 | 0
  Week 16 | 0
  Week 24 | 0
  Week 36 | 0
  Week 52 | 0

4. Secondary Outcome: Mean Change From Baseline in the Total GPP Score Over Time
Description: The Generalized Pustular Psoriasis (GPP) total score (range 0-17, with 17 representing severe disease) was calculated according to Japan Dermatology Association (JDA) severity index in GPP medical care guideline 2014. The total skin score (range 0-9, with 9 representing severe symptoms) is the combined skin scores for area of erythema (redness), area of erythema with pustules (small pockets of pus), and area of edema (swelling). The systemic and laboratory results score ([range 0-8, with 8 representing severe disease] assesses body temperature, white blood cell [WBC] count, high-sensitivity C-reactive protein [hs-CRP], and serum albumin). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
units on a scale
  Week 2 | -2.9 (2.08)
  Week 4 | -3.8 (2.15)
  Week 8 | -3.2 (2.57)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -3.1 (2.85)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -4.6 (1.85)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -3.8 (3.15)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -5.5 (2.07)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -6.0 (2.55)

5. Secondary Outcome: Mean Change From Baseline in JDA Severity Index of GPP Over Time
Description: The Generalized Pustular Psoriasis (GPP) total score (range 0-17, with 17 representing severe disease) was calculated according to Japan Dermatology Association (JDA) severity index in GPP medical care guideline 2014. The total skin score (range 0-9, with 9 representing severe symptoms) is the combined skin scores for area of erythema (redness), area of erythema with pustules (small pockets of pus), and area of edema (swelling). The systemic and laboratory results score ([range 0-8, with 8 representing severe disease] assesses body temperature, white blood cell [WBC] count, high-sensitivity C-reactive protein [hs-CRP], and serum albumin). A total score on the JDA severity index of 0-6 is categorized as "Mild", "Moderate" is 7-10, and "Severe" is 11-17.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Baseline: Mild | 3
  Baseline: Moderate | 6
  Baseline: Severe | 1
  Baseline: Missing | 0
  Week 2: Mild | 7
  Week 2: Moderate | 3
  Week 2: Severe | 0
  Week 2: Missing | 0
  Week 4: Mild | 9
  Week 4: Moderate | 1
  Week 4: Severe | 0
  Week 4: Missing | 0
  Week 8: Mild | 8
  Week 8: Moderate | 1
  Week 8: Severe | 1
  Week 8: Missing | 0
  Week 12: Mild | 7
  Week 12: Moderate | 0
  Week 12: Severe | 1
  Week 12: Missing | 2
  Week 16: Mild | 7
  Week 16: Moderate | 1
  Week 16: Severe | 0
  Week 16: Missing | 2
  Week 24: Mild | 7
  Week 24: Moderate | 0
  Week 24: Severe | 1
  Week 24: Missing | 2
  Week 36: Mild | 6
  Week 36: Moderate | 0
  Week 36: Severe | 0
  Week 36: Missing | 4
  Week 52: Mild | 5
  Week 52: Moderate | 0
  Week 52: Severe | 0
  Week 52: Missing | 5

6. Secondary Outcome: Mean Change From Baseline in Total Skin Score Over Time
Description: The Generalized Pustular Psoriasis (GPP) total skin score (range 0-9, with 9 representing severe symptoms) was calculated according to Japan Dermatology Association (JDA) severity index in GPP medical care guideline 2014. The total skin score is the combined skin scores for area of erythema (redness), area of erythema with pustules (small pockets of pus), and area of edema (swelling). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
units on a scale
  Week 2 | -1.9 (1.66)
  Week 4 | -2.4 (1.65)
  Week 8 | -2.3 (1.49)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -2.3 (1.98)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -3.1 (1.36)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -2.6 (1.92)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -3.8 (1.47)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -4.2 (1.79)

7. Secondary Outcome: Mean Percent Change From Baseline in Total Skin Score Over Time
Description: as for outcome 6
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
percentage change from baseline
  Week 2 | -33.8 (27.71)
  Week 4 | -43.4 (27.28)
  Week 8 | -42.9 (27.12)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -39.9 (30.36)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -54.6 (20.77)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -46.6 (33.15)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -67.9 (13.58)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -72.3 (16.34)

8. Secondary Outcome: Mean Change From Baseline in Total Systemic/Laboratory Test Score Over Time
Description: The Generalized Pustular Psoriasis (GPP) total systemic/laboratory test score ([range 0-8, with 8 representing severe disease] assesses body temperature, white blood cell [WBC] count, high-sensitivity C-reactive protein [hs-CRP], and serum albumin). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
units on a scale
  Week 2 | -1.0 (1.05)
  Week 4 | -1.4 (0.97)
  Week 8 | -0.9 (1.45)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -0.9 (1.25)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -1.5 (1.20)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -1.1 (1.64)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -1.7 (1.21)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -1.8 (1.30)

9. Secondary Outcome: Mean Change From Baseline in Total Erythema Area Over Time
Description: The Generalized Pustular Psoriasis (GPP) skin score scores for the total area of erythema (redness) were calculated according to Japan Dermatology Association (JDA) severity index in GPP medical care guideline 2014. The total erythema area is evaluated on a scale of 0 (none) to 3 (severe), with the percentage of body surface area involvement defined as follows: severe ≥ 75%; moderate, ≥ 25% and < 75%; mild, < 25%); and none (0%). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
units on a scale
  Week 2 | -17.0 (20.08)
  Week 4 | -21.6 (22.81)
  Week 8 | -19.7 (26.62)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -23.0 (26.28)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -34.6 (27.30)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -27.6 (29.48)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -48.3 (27.72)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -44.6 (37.50)

10. Secondary Outcome: Mean Change From Baseline in Total Erythema Area With Pustules Over Time
Description: The Generalized Pustular Psoriasis (GPP) skin score scores for the total area of erythema with pustules (small pockets of pus) were calculated according to Japan Dermatology Association (JDA) severity index in GPP medical care guideline 2014. The total erythema area with pustules is evaluated on a scale of 0 (none) to 3 (severe), with the percentage of body surface area involvement defined as follows: severe ≥ 50%; moderate, ≥ 10% and < 50%; mild, < 10%); and none (0%). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
units on a scale
  Week 2 | -9.3 (8.96)
  Week 4 | -11.7 (9.01)
  Week 8 | -8.3 (11.42)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -8.3 (14.63)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -11.8 (10.65)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -7.1 (16.75)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -13.3 (12.44)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -14.8 (13.31)

11. Secondary Outcome: Mean Change From Baseline in Total Edema Area Over Time
Description: The Generalized Pustular Psoriasis (GPP) skin score scores for the total area of edema (swelling) were calculated according to Japan Dermatology Association (JDA) severity index in GPP medical care guideline 2014. The total area of edema is evaluated on a scale of 0 (none) to 3 (severe), with the percentage of body surface area involvement defined as follows: severe ≥ 50%; moderate, ≥ 10% and < 50%; mild, < 10%); and none (0%). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
units on a scale
  Week 2 | -9.1 (9.45)
  Week 4 | -12.8 (11.29)
  Week 8 | -12.4 (17.30)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -6.3 (31.96)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -15.4 (17.30)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -14.0 (17.72)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -21.2 (14.68)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -18.6 (14.31)

12. Secondary Outcome: Mean Change From Baseline in Body Temperature Over Time
Description: Body temperature (oral) was obtained at each visit prior to blood sampling.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
degrees Celsius
  Week 2 | -0.3 (0.68)
  Week 4 | -0.5 (0.52)
  Week 8 | -0.3 (0.50)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -0.1 (0.64)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -0.3 (0.50)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -0.5 (1.04)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -0.3 (0.86)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -0.1 (0.64)

13. Secondary Outcome: Mean Change From Baseline in White Blood Cell (WBC) Concentration Over Time
Description: Blood was drawn at each study visit, and white blood cell concentration was determined.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
cells/µL
  Week 2 | -1220.0 (1970.22)
  Week 4 | -1770.0 (2572.96)
  Week 8 | -810.0 (3104.28)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -1650.0 (2857.57)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -2562.5 (2960.18)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -1162.5 (4444.88)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -2550.0 (3229.09)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -2760.0 (2966.99)

14. Secondary Outcome: Mean Change From Baseline in High-Sensitivity C-Reactive Protein (Hs-CRP) Over Time
Description: Blood was drawn at each study visit, and high-sensitivity C-reactive protein (hs-CRP) concentration was determined.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
mg/dL
  Week 2 | -1.5 (4.12)
  Week 4 | -1.6 (4.05)
  Week 8 | -0.3 (5.97)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -1.7 (4.76)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -2.5 (4.06)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -1.5 (5.63)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -2.7 (5.02)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -3.8 (4.73)

15. Secondary Outcome: Mean Change From Baseline in Serum Albumin Over Time
Description: Blood was drawn at each study visit, and serum albumin concentration was determined.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
g/dL
  Week 2 | 0.0 (0.33)
  Week 4 | 0.1 (0.44)
  Week 8 | 0.1 (0.38)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -0.2 (0.59)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -0.0 (0.39)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -0.0 (0.26)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -0.1 (0.54)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -0.0 (0.43)

16. Secondary Outcome: Number of Participants Achieving "Mild" in the JDA Severity Index of Generalized Pustular Psoriasis (GPP) for Participants With "Moderate" or "Severe" at Baseline Over Time
Description: as for outcome 5
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Week 2: number analyzed (Participants) | 7
  Week 2 | 4
  Week 4: number analyzed (Participants) | 7
  Week 4 | 6
  Week 8: number analyzed (Participants) | 7
  Week 8 | 5
  Week 12: number analyzed (Participants) | 7
  Week 12 | 5
  Week 16: number analyzed (Participants) | 7
  Week 16 | 5
  Week 24: number analyzed (Participants) | 7
  Week 24 | 5
  Week 36: number analyzed (Participants) | 7
  Week 36 | 5
  Week 52: number analyzed (Participants) | 7
  Week 52 | 4

17. Secondary Outcome: Proportion of Participants Achieving Treatment Success in Physician's Global Assessment of Generalized Pustular Psoriasis (PGA-GPP) Over Time
Description: The Physician's Global Assessment of Generalized Pustular Psoriasis (PGA-GPP) is a 6-point scale used to measure the severity of skin disease at the time of the qualified investigator's evaluation of the participant. The degree of overall severity was evaluated using the following categories: erythema, pustulation, and edema, and graded as follows. Grade 0 = cleared, except for residual discoloration; Grade 1 = minimal; Grade 2 = mild; Grade 3 = moderate; Grade 4 = severe; and Grade 5 = very severe. The score is an arithmetic average of the grades for erythema, pustulation, and edema, rounded to the nearest whole number. Treatment Success was defined by at least a 2 grade improvement relative to baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Week 2 | 3
  Week 4 | 5
  Week 8 | 4
  Week 12: number analyzed (Participants) | 8
  Week 12 | 3
  Week 16: number analyzed (Participants) | 8
  Week 16 | 5
  Week 24: number analyzed (Participants) | 8
  Week 24 | 4
  Week 36: number analyzed (Participants) | 6
  Week 36 | 5
  Week 52: number analyzed (Participants) | 5
  Week 52 | 3

18. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Generalized Pustular Psoriasis (PGA-GPP) Grade Over Time
Description: The Physician's Global Assessment of Generalized Pustular Psoriasis (PGA-GPP) is a 6-point scale used to measure the severity of skin disease at the time of the qualified investigator's evaluation of the participant. The degree of overall severity was evaluated using the following categories: erythema, pustulation, and edema, and graded as follows. Grade 0 = cleared, except for residual discoloration; Grade 1 = minimal; Grade 2 = mild; Grade 3 = moderate; Grade 4 = severe; and Grade 5 = very severe. The score is an arithmetic average of the grades for erythema, pustulation, and edema, rounded to the nearest whole number.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Baseline: PGA Grade 0 | 0
  Baseline: PGA Grade 1 | 0
  Baseline: PGA Grade 2 | 4
  Baseline: PGA Grade 3 | 3
  Baseline: PGA Grade 4 | 3
  Baseline: PGA Grade 5 | 0
  Week 2: PGA Grade 0 | 1
  Week 2: PGA Grade 1 | 3
  Week 2: PGA Grade 2 | 5
  Week 2: PGA Grade 3 | 1
  Week 2: PGA Grade 4 | 0
  Week 2: PGA Grade 5 | 0
  Week 4: PGA Grade 0 | 1
  Week 4: PGA Grade 1 | 7
  Week 4: PGA Grade 2 | 1
  Week 4: PGA Grade 3 | 1
  Week 4: PGA Grade 4 | 0
  Week 4: PGA Grade 5 | 0
  Week 8: PGA Grade 0 | 0
  Week 8: PGA Grade 1 | 8
  Week 8: PGA Grade 2 | 0
  Week 8: PGA Grade 3 | 1
  Week 8: PGA Grade 4 | 1
  Week 8: PGA Grade 5 | 0
  Week 12: number analyzed (Participants) | 8
  Week 12: PGA Grade 0 | 1
  Week 12: PGA Grade 1 | 4
  Week 12: PGA Grade 2 | 2
  Week 12: PGA Grade 3 | 0
  Week 12: PGA Grade 4 | 0
  Week 12: PGA Grade 5 | 1
  Week 16: number analyzed (Participants) | 8
  Week 16: PGA Grade 0 | 2
  Week 16: PGA Grade 1 | 5
  Week 16: PGA Grade 2 | 1
  Week 16: PGA Grade 3 | 0
  Week 16: PGA Grade 4 | 0
  Week 16: PGA Grade 5 | 0
  Week 24: number analyzed (Participants) | 8
  Week 24: PGA Grade 0 | 1
  Week 24: PGA Grade 1 | 5
  Week 24: PGA Grade 2 | 0
  Week 24: PGA Grade 3 | 2
  Week 24: PGA Grade 4 | 0
  Week 24: PGA Grade 5 | 0
  Week 36: number analyzed (Participants) | 6
  Week 36: PGA Grade 0 | 2
  Week 36: PGA Grade 1 | 4
  Week 36: PGA Grade 2 | 0
  Week 36: PGA Grade 3 | 0
  Week 36: PGA Grade 4 | 0
  Week 36: PGA Grade 5 | 0
  Week 52: number analyzed (Participants) | 5
  Week 52: PGA Grade 0 | 3
  Week 52: PGA Grade 1 | 2
  Week 52: PGA Grade 2 | 0
  Week 52: PGA Grade 3 | 0
  Week 52: PGA Grade 4 | 0
  Week 52: PGA Grade 5 | 0

19. Secondary Outcome: Proportion of Participants Achieving Physician's Global Assessment of Generalized Pustular Psoriasis (PGA-GPP) Grade 0 or 1 for Those With PGA Grade of at Least 2 at Baseline Over Time
Description: as for outcome 18
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Week 2 | 4
  Week 4 | 8
  Week 8 | 8
  Week 12: number analyzed (Participants) | 8
  Week 12 | 5
  Week 16: number analyzed (Participants) | 8
  Week 16 | 7
  Week 24: number analyzed (Participants) | 8
  Week 24 | 6
  Week 36: number analyzed (Participants) | 6
  Week 36 | 6
  Week 52: number analyzed (Participants) | 5
  Week 52 | 5

20. Secondary Outcome: Proportion of Participants Achieving Psoriasis Area and Severity Index 90 (PASI 90) Over Time
Description: The proportion of participants with a ≥ 90% reduction (improvement) in the Psoriasis Area and Severity Index (PASI) score from baseline was calculated. PASI is a combination of the intensity of psoriasis, assessed for erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Week 2 | 1
  Week 4 | 2
  Week 8 | 1
  Week 12: number analyzed (Participants) | 8
  Week 12 | 1
  Week 16: number analyzed (Participants) | 8
  Week 16 | 0
  Week 24: number analyzed (Participants) | 8
  Week 24 | 1
  Week 36: number analyzed (Participants) | 6
  Week 36 | 3
  Week 52: number analyzed (Participants) | 5
  Week 52 | 3

21. Secondary Outcome: Proportion of Participants Achieving Psoriasis Area and Severity Index 75 (PASI 75) Over Time
Description: The proportion of participants with a ≥ 75% reduction (improvement) in the Psoriasis Area and Severity Index (PASI) score from baseline was calculated. PASI is a combination of the intensity of psoriasis, assessed for erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Week 2 | 2
  Week 4 | 2
  Week 8 | 2
  Week 12: number analyzed (Participants) | 8
  Week 12 | 2
  Week 16: number analyzed (Participants) | 8
  Week 16 | 4
  Week 24: number analyzed (Participants) | 8
  Week 24 | 4
  Week 36: number analyzed (Participants) | 6
  Week 36 | 5
  Week 52: number analyzed (Participants) | 5
  Week 52 | 3

22. Secondary Outcome: Proportion of Participants Achieving Psoriasis Area and Severity Index 50 (PASI 50) Over Time
Description: The proportion of participants with a ≥ 50% reduction (improvement) in the Psoriasis Area and Severity Index (PASI) score from baseline was calculated. PASI is a combination of the intensity of psoriasis, assessed for erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Week 2 | 4
  Week 4 | 6
  Week 8 | 6
  Week 12: number analyzed (Participants) | 8
  Week 12 | 5
  Week 16: number analyzed (Participants) | 8
  Week 16 | 5
  Week 24: number analyzed (Participants) | 8
  Week 24 | 4
  Week 36: number analyzed (Participants) | 6
  Week 36 | 5
  Week 52: number analyzed (Participants) | 5
  Week 52 | 4

23. Secondary Outcome: Mean Change From Baseline in Psoriasis Area and Severity Index (PASI) Score Over Time
Description: The mean change in the Psoriasis Area and Severity Index (PASI) score from baseline was calculated. PASI is a combination of the intensity of psoriasis, assessed for erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
units on a scale
  Week 2 | -12.9 (12.83)
  Week 4 | -17.4 (14.66)
  Week 8 | -14.9 (17.55)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -14.3 (20.03)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -19.1 (17.27)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -16.8 (19.61)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -28.1 (17.67)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -26.7 (22.24)

24. Secondary Outcome: Mean Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score Over Time
Description: The percent change in the Psoriasis Area and Severity Index (PASI) score from baseline was calculated. PASI is a combination of the intensity of psoriasis, assessed for erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
percentage change from baseline
  Week 2 | -44.2 (27.47)
  Week 4 | -59.7 (24.65)
  Week 8 | -43.9 (45.01)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -45.0 (39.20)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -55.5 (31.89)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -43.6 (46.26)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -79.0 (24.13)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -33.7 (117.4)

25. Secondary Outcome: Proportion of Participants Achieving Dermatology Life Quality Index (DLQI) Score of 0 Over Time
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment- related feelings. Participants respond to 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means that psoriasis has an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all.
Time Frame: Week 8, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Week 8 | 1
  Week 16: number analyzed (Participants) | 8
  Week 16 | 0
  Week 24: number analyzed (Participants) | 8
  Week 24 | 1
  Week 36: number analyzed (Participants) | 6
  Week 36 | 0
  Week 52: number analyzed (Participants) | 5
  Week 52 | 2

26. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI) Score Over Time
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment- related feelings. Participants respond to 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means that psoriasis has an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 8, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
units on a scale
  Week 8 | -4.2 (6.55)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -6.6 (5.34)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -4.8 (7.59)
  Week 36: number analyzed (Participants) | 6
  Week 36 | -6.5 (5.65)
  Week 52: number analyzed (Participants) | 5
  Week 52 | -8.0 (7.18)

27. Secondary Outcome: Mean Change From Baseline in Short Form-36 Health Status Survey Version 2 (SF-36 V2) Score Over Time
Description: The Short Form-36 Health Status Survey Version 2 (SF-36 V2) is a 36-item generic health-related quality of life questionnaire to assess the participant's view of their health consisting of 2 components: physical and mental. For each component, a transformed summary score is calculated using 8 sub-domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 100. Higher scores indicate a better health state.
Time Frame: Baseline, Week 8, Week 16, Week 24, Week 36, Week 52
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
units on a scale
  Physical Component Summary- Week 8 | 4.7 (19.05)
  Physical Component Summary- Week 16: number analyzed (Participants) | 8
  Physical Component Summary- Week 16 | 9.2 (17.48)
  Physical Component Summary- Week 24: number analyzed (Participants) | 8
  Physical Component Summary- Week 24 | 8.2 (15.94)
  Physical Component Summary- Week 36: number analyzed (Participants) | 6
  Physical Component Summary- Week 36 | 4.9 (23.39)
  Physical Component Summary- Week 52: number analyzed (Participants) | 5
  Physical Component Summary- Week 52 | 12.0 (21.42)
  Mental Component Summary- Week 8 | 0.6 (8.71)
  Mental Component Summary- Week 16: number analyzed (Participants) | 8
  Mental Component Summary- Week 16 | 0.9 (8.03)
  Mental Component Summary- Week 24: number analyzed (Participants) | 8
  Mental Component Summary- Week 24 | 2.0 (8.32)
  Mental Component Summary- Week 36: number analyzed (Participants) | 6
  Mental Component Summary- Week 36 | 1.6 (18.26)
  Mental Component Summary- Week 52: number analyzed (Participants) | 5
  Mental Component Summary- Week 52 | 6.4 (7.79)

28. Secondary Outcome: Proportion of Participants Taking Systemic Co-medication for Generalized Pustular Psoriasis (GPP) at Any Time During the Study
Description: GPP-specific co-medications were documented at each scheduled study visit.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Etretinate | 3
  Methotrexate | 2
  Oral steroids | 1
  Cyclosporine | 2

29. Secondary Outcome: Proportion of Participants Taking Topical Co-medication for Generalized Pustular Psoriasis (GPP) at Any Time During the Study
Description: Participants using topical co-medications for GPP were documented at each scheduled study visit.
Time Frame: as for outcome 28
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 10
Participants
  Corticosteroid | 7
  Vitamin D3 | 0
  Tacrolimus | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 70 days after the last dose of study drug (up to 62 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 70 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Participants Receiving Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Adalimumab (N=10)
Cardiac failure (Cardiac disorders) | 1
Chronic sinusitis (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Adalimumab (N=10)
Eosinophilia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Autoimmune Thyroiditis (Endocrine disorders) | 1
Dry eye (Eye disorders) | 1
Episcleritis (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Hepatic Steatosis (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Bacterial infection (Infections and infestations) | 1
Body tinea (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Eye contusion (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Insomnia (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT02533375/SAP_000.pdf
  • Study Protocol (2015-06-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT02533375/Prot_001.pdf